CLINICAL TRIAL: NCT06260202
Title: Nutrition Under Noninvasive Ventilation in Critically Ill Patients: a Retrospective Monocentric Analysis
Brief Title: Nutrition Under Noninvasive Ventilation
Acronym: NUTRINIV
Status: Completed | Type: Observational
Sponsor: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Responsible Party: Principal Investigator, Francesca Moretto, Principal Investigator, Università degli Studi del Piemonte Orientale Amedeo Avogadro
Other Study IDs: 308.273
Record Dates: First submitted 2024-01-29; First posted 2024-02-15 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Noninvasive Ventilation; Nutrition Therapy; Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Even though nutrition is a fundamental component of Intensive care unit (ICU) therapy, critically ill patients are frequently malnourished, a factor well known for its strong association with a higher risk of complications, prolonged ICU/hospital length of stay, and greater ICU readmission and mortality rates. Noninvasive ventilation (NIV) use has increased considerably over the past twenty years, making this supportive technique a keystone of acute respiratory failure (ARF) treatment. In this setting, respiratory support is provided through an interface, usually a mask or a helmet, that frequently represents an important obstacle to nutrition delivery, making oral intake impossible and posing the necessity to start enteral (EN) or parenteral nutrition (PN). Moreover, while critical care guidelines regarding nutritional management of patients receiving mechanical ventilation (MV) are well established, data and recommendations about the appropriate nutritional support to patients in NIV are still very limited. Due to this limited data, we want to describe characteristics and nutritional management of patients undergoing NIV in ICU, and to evaluate the difference between the mean caloric and protein intake of these patients and the recommended caloric and protein target for critically ill patients. Secondarily, we want to evaluate the difference of the caloric and protein intake among groups of patients undergoing different nutritional modality and to assess potential associations of the nutritional characteristics with patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients;
* Admission to the Intensive Care Unit of Maggiore della Carità University Hospital from March 1st 2020 to February 28th 2023;
* Noninvasive ventilation treatment for acute respiratory failure of any cause;
* Duration of noninvasive ventilation treatment of more than two days;
* Informed consent signed.

Exclusion Criteria:

* Patients under 18 years of age;
* Duration of noninvasive ventilation treatment of less than two days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the Intensive Care Unit of Maggiore della Carità University Hospital from March 1st 2020 to February 28th 2023, undergoing noninvasive ventilation for any diagnosis of acute respiratory failure and for any cause (to avoid endotracheal intubation, as alternative to invasive ventilation, as weaning from invasive ventilation) will be considered.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Caloric and protein gap | At ICU discharge, a median of six days
  to evaluate the difference between the mean caloric and protein intake of these patients and the recommended caloric and protein target for critically ill patients for every day of ICU stay

SECONDARY OUTCOMES:
Nutrition modalities outcomes | At ICU discharge, a median of six days
  to evaluate the difference of the mean caloric and protein intake among groups of patients undergoing different nutritional modality

CONTACTS AND LOCATIONS:
Locations (1):
- Università del Piemonte Orientale, Novara, Italy